CLINICAL TRIAL: NCT02693054
Title: Characterizing Safety and Efficacy of Halo Hybrid Fractional Laser Treatments for Various Skin Conditions
Brief Title: Safety and Efficacy Study for Various Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HALOCIP001
Record Dates: First submitted 2016-02-08; First posted 2016-02-26 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Dyschromia; Photodamaged Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hybrid Fractional Laser Treatment (Experimental): Halo (1470nm and 2940 nm) laser
  Interventions: Device: HALO

INTERVENTIONS:
Device: HALO — Laser Treatment

SUMMARY:
Characterizing safety and efficacy of Halo Laser Treatment for Various Skin Conditions.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate safety and efficacy of Halo treatment as measured by changes in skin tone, texture and pigment.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin types I to IV
* Desires improvement of significant skin conditions on the face and/or neck
* Willingness to participate in the study by signing an informed consent form
* Will have limited sun exposure for at least two weeks prior to study screening and during the study, including the follow-up period
* Able to adhere to the treatment and follow-up schedule and post-treatment care instructions
* Post-menopausal or surgically sterilized female subjects.

Exclusion Criteria:

* History of Halo or resurfacing procedures in the treatment area within past six months
* Has tanned within the past thirty days or unable or unlikely to refrain from tanning, including the use of tanning booths, tanning spray, or cream
* Has tattoos, dysplastic nevi in the treatment area
* Pregnant and/or lactating
* Is planning to get pregnant within the study period
* Has a known history of photosensitivity
* Has used medication with photosensitizing properties within the past six months, e.g. isotretinoin
* History or evidence of chronic or recurring skin disease or disorder (e.g. psoriasis, --Netherton syndrome, etc.) affecting the treatment area
* Has open lacerations, abrasions, active cold sores, or herpes sores
* Has hormonal disorders
* History of keloid or hypertrophic scar formation or poor wound healing
* History of immunosuppression or immune deficiency disorder (including HIV infection or AIDS) or use of immunosuppressive medications
* History of bleeding disorder or taking anticoagulation medications
* History of skin cancer or any other cancer in the treatment area
* Has significant concurrent illnesses, such as diabetes, lupus, epilepsy, or cardiac disorders, which might be aggravated as a result of treatment
* Has participated in any clinical trial involving an investigational drug or cosmetic product or procedure within the past thirty days
* The investigator feels that for any reason the subject is not eligible to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement in skin conditions assessed by photographs | 6 months
  Assessment of photographs by blinded evaluators

SECONDARY OUTCOMES:
Subject satisfaction post final treatment | 3 months
  Assessment of subject satisfaction with treatment result using survey/questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jason Pozner, MD, Principal Investigator — Sanctuary Plastic Surgery; Christopher Robb, MD, Principal Investigator — Skin and Allergy Center; Elizabeth Tanzi, MD, Principal Investigator — Capital Laser and Skin Care; Jill Waibel, MD, Principal Investigator — Miami Dermatology and Laser Institute

IPD SHARING:
Plan to Share IPD: No